CLINICAL TRIAL: NCT04319003
Title: Surveillance of Obesity and Pre-Diabetes/Diabetes in Kiritimati School Children and Lifestyle Modifications to Reduce Risk
Brief Title: Pilot Sugar Reduction Intervention in Kiritimati Teenagers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Elizabeth Beale, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS-18-00505
Record Dates: First submitted 2020-02-26; First posted 2020-03-24 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control School (No Intervention): This school did not receive intervention (until after the study was completed)
- Intervention School (Experimental): This school received a one-week sugar-reduction intervention
  Interventions: Behavioral: Sugar-reduction intervention

INTERVENTIONS:
Behavioral: Sugar-reduction intervention — The intervention consisted of a) installation of a water filter at the school. b) each participant received a metal water bottle. c) a registered dietitian gave a 30-minute presentation on sugar reduction for the purposes of type 2 diabetes prevention
  Arms: Intervention School

SUMMARY:
Kiritimati is an isolated coral atoll in the Pacific Ocean, and is one of 32 islands that comprise the Republic of Kiribati. Obesity and type 2 diabetes rates are high in Kiribati, but the causes and rates of childhood obesity/diabetes are unknown. However, it has been hypothesized that high consumption of sugar-sweetened beverages on Kiritimati may be a contributing factor. The investigators therefore conducted a study in Kiritimati in September 2018 with the aim of 1) quantifying obesity and diabetes rates amongst children on Kiritimati and 2) testing the feasibility of a sugar-reduction intervention in Kiritimati schools. The investigators randomized the two high schools on the island to either the control group or the intervention group. The investigators measured height/weight, continuous blood glucose (using flash glucose monitoring), and diet (using 24-hour diet recalls). One week into the study, the intervention school received an intervention, which consisted of installation of a water filter at the school, the provision of water bottles to each student at the school, and a 30-minute educational presentation on the link between sugar consumption and type 2 diabetes. The investigators then measured how blood glucose and diet changed the week following the intervention, and compared this to the control school.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in one of the two high schools on Kiritimati

Exclusion Criteria:

* > 18 years of age

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

PRIMARY OUTCOMES:
Change in mean blood glucose (mg/dL) | 2 weeks (1 week pre- and 1 week post-intervention)
  A continuous glucose monitor was attached to all participants, which collected data for 2 weeks. Mean blood glucose was calculated for each participant using GlyCulator, an online tool for analyzing CGM data.
Change in mean amplitude of glycemic variability (MAGE) (mg/dL) | 2 weeks (1 week pre- and 1 week post-intervention)
  A continuous glucose monitor was attached to all participants, which collected data for 2 weeks. Glycemic variability (mean amplitude of glycemic excursions) was calculated for each participant using GlyCulator, an online tool for analyzing CGM data.
Change in standard deviation (mg/dL) of continuous glucose monitor data | 2 weeks (1 week pre- and 1 week post-intervention)
  A continuous glucose monitor was attached to all participants, which collected data for 2 weeks. Glycemic variability (standard deviation) was calculated for each participant using GlyCulator, an online tool for analyzing CGM data.
Change in coefficient of variation (percent) of continuous glucose monitor data | 2 weeks (1 week pre- and 1 week post-intervention)
  A continuous glucose monitor was attached to all participants, which collected data for 2 weeks. Glycemic variability (coefficient of variation (percent) was calculated for each participant using GlyCulator, an online tool for analyzing CGM data.
Change in J-index of continuous glucose monitor data | 2 weeks (1 week pre- and 1 week post-intervention)
  A continuous glucose monitor was attached to all participants, which collected data for 2 weeks. Glycemic variability (J-index) was calculated for each participant using GlyCulator, an online tool for analyzing CGM data.
Change in area under the curve of continuous glucose monitor data | 2 weeks (1 week pre- and 1 week post-intervention)
  A continuous glucose monitor was attached to all participants, which collected data for 2 weeks. Glycemic variability (area under the curve) was calculated for each participant using GlyCulator, an online tool for analyzing CGM data.
Change in total sugar consumption (g/day) using 24-hour dietary recalls | 2 weeks (1 week pre- and 1 week post-intervention)
  The investigators conducted 24-hour diet recalls and entered data into the NDSR database for comparison of change in total sugar intake between the control and intervention schools (time x group interaction).
Change in added sugar consumption (g/day) using 24-hour dietary recalls | 2 weeks (1 week pre- and 1 week post-intervention)
  The investigators conducted 24-hour diet recalls and entered data into the NDSR database for comparison of change in added sugar intake between the control and intervention schools (time x group interaction).
Change in total water consumption (g/day) using 24-hour dietary recalls | 2 weeks (1 week pre- and 1 week post-intervention)
  The investigators conducted 24-hour diet recalls and entered data into the NDSR database for comparison of change in total water intake between the control and intervention schools (time x group interaction).
Change in unsweetened water consumption (servings/day) using 24-hour dietary recalls | 2 weeks (1 week pre- and 1 week post-intervention)
  The investigators conducted 24-hour diet recalls and entered data into the NDSR database for comparison of change in unsweetened water intake between the control and intervention schools (time x group interaction).
Change in energy (kcal/day) consumption using 24-hour dietary recalls | 2 weeks (1 week pre- and 1 week post-intervention)
  The investigators conducted 24-hour diet recalls and entered data into the NDSR database for comparison of change in energy (kcal) intake between the control and intervention schools (time x group interaction).
Change in total carbohydrate (g/day) consumption using 24-hour dietary recalls | 2 weeks (1 week pre- and 1 week post-intervention)
  The investigators conducted 24-hour diet recalls and entered data into the NDSR database for comparison of change in total carbohydrate intake between the control and intervention schools (time x group interaction).
Change in percent calories from carbohydrate consumption using 24-hour dietary recalls | 2 weeks (1 week pre- and 1 week post-intervention)
  The investigators conducted 24-hour diet recalls and entered data into the NDSR database for comparison of change in % calories from carbohydrate intake between the control and intervention schools (time x group interaction).
Change in percent calories from total sugars consumption using 24-hour dietary recalls | 2 weeks (1 week pre- and 1 week post-intervention)
  The investigators conducted 24-hour diet recalls and entered data into the NDSR database for comparison of change in % calories from total sugars intake between the control and intervention schools (time x group interaction).
Change in percent calories from added sugars consumption using 24-hour dietary recalls | 2 weeks (1 week pre- and 1 week post-intervention)
  The investigators conducted 24-hour diet recalls and entered data into the NDSR database for comparison of change in % calories from added sugars intake between the control and intervention schools (time x group interaction).
Change in sugary beverage (tioka) consumption using beverage frequency questionnaires | 2 weeks (1 week pre- and 1 week post-intervention)
  The investigators conducted beverage frequency questionnaires which asked about consumption of popular beverages on Kiritimati (specifically: "how many days per week do you typically drink this drink?" and "how much each day?") then compared change pre-and post-intervention between the two groups (time x group interaction) in servings/day.
Change in sugary beverage (tang) consumption using beverage frequency questionnaires | 2 weeks (1 week pre- and 1 week post-intervention)
  The investigators conducted beverage frequency questionnaires which asked about consumption of popular beverages on Kiritimati (specifically: "how many days per week do you typically drink this drink?" and "how much each day?") then compared change pre-and post-intervention between the two groups (time x group interaction) in servings/day.
Change in sugary beverage (toddy) consumption using beverage frequency questionnaires | 2 weeks (1 week pre- and 1 week post-intervention)
  The investigators conducted beverage frequency questionnaires which asked about consumption of popular beverages on Kiritimati (specifically: "how many days per week do you typically drink this drink?" and "how much each day?") then compared change pre-and post-intervention between the two groups (time x group interaction) in servings/day.
Change in sugary beverage (ice block) consumption using beverage frequency questionnaires | 2 weeks (1 week pre- and 1 week post-intervention)
  The investigators conducted beverage frequency questionnaires which asked about consumption of popular beverages on Kiritimati (specifically: "how many days per week do you typically drink this drink?" and "how much each day?") then compared change pre-and post-intervention between the two groups (time x group interaction) in servings/day.
Change in sugary beverage (soda) consumption using beverage frequency questionnaires | 2 weeks (1 week pre- and 1 week post-intervention)
  The investigators conducted beverage frequency questionnaires which asked about consumption of popular beverages on Kiritimati (specifically: "how many days per week do you typically drink this drink?" and "how much each day?") then compared change pre-and post-intervention between the two groups (time x group interaction) in servings/day.
Change in sugary beverage (juice) consumption using beverage frequency questionnaires | 2 weeks (1 week pre- and 1 week post-intervention)
  The investigators conducted beverage frequency questionnaires which asked about consumption of popular beverages on Kiritimati (specifically: "how many days per week do you typically drink this drink?" and "how much each day?") then compared change pre-and post-intervention between the two groups (time x group interaction) in servings/day.
Change in sugary beverage (fruit drinks) consumption using beverage frequency questionnaires | 2 weeks (1 week pre- and 1 week post-intervention)
  The investigators conducted beverage frequency questionnaires which asked about consumption of popular beverages on Kiritimati (specifically: "how many days per week do you typically drink this drink?" and "how much each day?") then compared change pre-and post-intervention between the two groups (time x group interaction) in servings/day.
Change in sugary beverage (coffee/tea) consumption using beverage frequency questionnaires | 2 weeks (1 week pre- and 1 week post-intervention)
  The investigators conducted beverage frequency questionnaires which asked about consumption of popular beverages on Kiritimati (specifically: "how many days per week do you typically drink this drink?" and "how much each day?") then compared change pre-and post-intervention between the two groups (time x group interaction) in servings/day.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Beale, MD, Principal Investigator — University of Southern California
Locations (2):
- University of Southern California, Los Angeles, California, United States
- Kiritimati, London, Kiribati

IPD SHARING:
Plan to Share IPD: No